CLINICAL TRIAL: NCT05783102
Title: Knowledge and Interpersonal Skills to Develop Exemplary Relationships (Pilot 2)
Brief Title: Knowledge and Interpersonal Skills to Develop Exemplary Relationships (KINDER): Pilot Study
Acronym: KINDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Kylie Meyer, Assistant Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20221333
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Caregiver Burden; Relation, Family; Elder Abuse
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KINDER Intervention (Experimental): KINDER is a 9-week psychoeducational intervention.
  Interventions: Behavioral: Knowledge and Interpersonal Skills to Develop Exemplary Relationships

INTERVENTIONS:
Behavioral: Knowledge and Interpersonal Skills to Develop Exemplary Relationships — During this 9-week psychoeducational intervention, participants will complete eight weekly, self-paced lessons that include a short video vignette, written text, a reading quiz, and a reflection exercise. Topics include understanding a dementia diagnosis, communicating with a person you care for about challenging topics, finding a balance between safety concerns and independence, and more. Each lesson takes an estimated 1 hour to complete. Independent KINDER lessons can be completed using a printed or digital copy of the KINDER Workbook. In addition, participants will be asked to participate in three, 1.5-hour group discussion sessions with other caregivers and a facilitator. These sessions will take place over Zoom video conference.

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of delivering the KINDER intervention to family caregivers to persons living with dementia. Further, the investigators will examine the preliminary efficacy of the KINDER intervention at improving caregiver resourcefulness, relationship quality, and quality of care, including reduction of potential verbal-type elder mistreatment.

During this study, participants will be asked to complete two (2) 30- to 45-minute surveys asking about their demographic information, caregiving situations, and relationship with the care recipient. The first survey will be sent within two weeks of beginning the KINDER intervention, the second will be sent within one week after participants complete the KINDER intervention so we can compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Is age 18+
* Provides care to a family member or friend living with Alzheimer's Disease or a related dementia.
* Helps with at least 1 activity of daily living (e.g., bathing) or 2 instrumental activities of daily living (e.g., shopping)
* Provides at least 8 hours of assistance to the care recipient per week
* Does not intend to place the care recipient in a skilled nursing facility within 3 months of consenting into the study

Exclusion Criteria:

* Does not read and speak English
* Cannot reliably access a computer and internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kylie N Meyer, PhD, MSc, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acierno R, Hernandez MA, Amstadter AB, Resnick HS, Steve K, Muzzy W, Kilpatrick DG. Prevalence and correlates of emotional, physical, sexual, and financial abuse and potential neglect in the United States: the National Elder Mistreatment Study. Am J Public Health. 2010 Feb;100(2):292-7. doi: 10.2105/AJPH.2009.163089. Epub 2009 Dec 17. PMID 20019303
- [Background] Burnes D, Pillemer K, Lachs MS. Elder Abuse Severity: A Critical but Understudied Dimension of Victimization for Clinicians and Researchers. Gerontologist. 2017 Aug 1;57(4):745-756. doi: 10.1093/geront/gnv688. PMID 26874186
- [Background] Conrad KJ, Iris M, Ridings JW, Langley K, Anetzberger GJ. Self-report measure of psychological abuse of older adults. Gerontologist. 2011 Jun;51(3):354-66. doi: 10.1093/geront/gnq103. Epub 2010 Dec 20. PMID 21173437
- [Background] DeLiema M, Gassoumis ZD, Homeier DC, Wilber KH. Determining prevalence and correlates of elder abuse using promotores: low-income immigrant Latinos report high rates of abuse and neglect. J Am Geriatr Soc. 2012 Jul;60(7):1333-9. doi: 10.1111/j.1532-5415.2012.04025.x. Epub 2012 Jun 14. PMID 22697790
- [Background] Gitlin LN, Winter L, Dennis MP, Corcoran M, Schinfeld S, Hauck WW. Strategies used by families to simplify tasks for individuals with Alzheimer's disease and related disorders: psychometric analysis of the Task Management Strategy Index (TMSI). Gerontologist. 2002 Feb;42(1):61-9. doi: 10.1093/geront/42.1.61. PMID 11815700
- [Background] McClendon MJ, Smyth KA. Quality of informal care for persons with dementia: dimensions and correlates. Aging Ment Health. 2013;17(8):1003-15. doi: 10.1080/13607863.2013.805400. Epub 2013 Jun 11. PMID 24171485
- [Background] Reamy AM, Kim K, Zarit SH, Whitlatch CJ. Understanding discrepancy in perceptions of values: individuals with mild to moderate dementia and their family caregivers. Gerontologist. 2011 Aug;51(4):473-83. doi: 10.1093/geront/gnr010. Epub 2011 Mar 7. PMID 21383111
- [Background] Straus, MA, Hamby, SL, Boney-McCoy, SUE, & Sugarman, DB. The Revised Conflict Tactics Scales (CTS2). Journal of Family Issues. 2016; 17(3): 283-316. doi: 10.1177/01925139601700300.
- [Background] Zauszniewski JA, Lai CY, Tithiphontumrong S. Development and testing of the Resourcefulness Scale for Older Adults. J Nurs Meas. 2006 Spring-Summer;14(1):57-68. doi: 10.1891/jnum.14.1.57. PMID 16764178
- [Derived] Meyer K, Wei W, Yonashiro-Cho J, Mage S, Kim S, Irani E, Burant C, Gassoumis Z, Lamb EG, Zauszniewski JA, Benton D. Acceptability of an Intervention to Prevent Older Adult Mistreatment Among Family Caregivers to Persons With Dementia: Multimethod Pilot Study. JMIR Form Res. 2025 Jul 30;9:e73778. doi: 10.2196/73778. PMID 40737062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KINDER Intervention
Started | 45
Completed | 42
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | KINDER Intervention
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants had missing data for this variable.
  years
    number analyzed (Participants) | 43
    (all) | 58.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant had missing data for this variable.
  Participants
    number analyzed (Participants) | 44
    Female | 39
    Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 5
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Resourcefulness
Description: Resourcefulness is measured using the 28-item Caregiver Resourcefulness Scale (α=0.85; Zauszniewski, 2006). This scale has two factors: one focused on help-seeking and another on self-help. Caregivers are asked the frequency at which they use different strategies to manage challenges, and may respond: Not at all like me (0), Pretty much not like me (1), A little bit not like me (2), A little bit like me (3), Pretty much like much like me (4), or Very much like me (5). Items are added together to create a total score. Scores range from 0 to 140, where higher scores indicate higher levels of resourcefulness. The outcome measure will use the average change score from baseline scores until the post-intervention survey.
Time Frame: Change from baseline to post-intervention (within 2 weeks after the 9 weeks intervention).
Population: Only participants who completed the Caregiver Resourcefulness Scale without missing data were included in the analysis. This explains why the number of participants analyzed is lower than the overall total number of study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KINDER Intervention
Number analyzed (Participants) | 28
score on a scale | 9.20 (14.3)

2. Secondary Outcome: Caregiving Relationship Strain
Description: Relationship strain will be measured using the 5-item Strain Scale of the Dyadic Relationship Scale (α=0.69; Reamy et al., 2011). Respondents are asked to indicate agreement with statements such as, "The patient made too many requests," and may indicate Strongly Disagree, Disagree, Agree, or Strongly Agree. The scale has a range of scores from 4 to 20, where higher scores indicate greater levels of relationship strain. The outcome measure will use the average change score from baseline scores until the post-intervention survey.
Time Frame: Change from baseline to post-intervention (within 2 weeks after the 9 weeks intervention).
Population: Only participants who completed the Caregiving Relationship Scale without missing data were included in the analysis. This explains why the number of participants analyzed is lower than the overall total number of study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KINDER Intervention
Number analyzed (Participants) | 34
score on a scale | -2.6 (3.3)

3. Secondary Outcome: Quality of Caregiving
Description: Quality of caregiving will be measured with the Task Management Strategy Index (TMSI; α=0.74 to 0.81; McClendon & Smyth, 2013). The 19-item TMSI was developed to assess caregivers' ability to manage their family member's functional disabilities. (Gitlin et al., 2002) Caregivers are asked how often they engage in strategies that support quality care. Caregivers indicate Never, Rarely, Sometimes, Often, or Always. Scores range from 19 to 95. Higher scores indicate higher quality of caregiving. The outcome measure will use the average change score from baseline scores until the post-intervention survey.
Time Frame: Change from baseline to post-intervention (within 2 weeks after the 9 weeks intervention).
Population: Only participants who completed the Quality of Caregiving Scale without missing data were included in the analysis. This explains why the number of participants analyzed is lower than the overall total number of study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KINDER Intervention
Number analyzed (Participants) | 26
score on a scale | 6.0 (13.7)

4. Secondary Outcome: Frequency of Psychological Elder Mistreatment
Description: The investigators will use a modified version of the Conflict Tactics Scale 2 to measure psychological elder mistreatment (MCTS 2; α=0.79; Straus et al., 2016). Items include behaviors such as insulting, swearing at, or yelling at a partner. To measure a range of psychological elder mistreatment behaviors, we will add three items: ignoring the care recipient (DeLiema et al., 2012), threatening to isolate the care recipient (Acierno et al., 2010), and talking about the care recipient as if they are not there (Conrad et al., 2011). To describe the severity of mistreatment (Burnes et al., 2017), participants will be asked to describe the frequency of each behavior, such that response options will include: None, Once, Twice, 3 to 5 times, 6 to 10 times, and More than 10 times. Scores range from 0 to 50. Higher scores indicate higher quality of caregiving. The outcome measure will use the average change score from baseline scores until the post-intervention survey.
Time Frame: Change from baseline to post-intervention (within 2 weeks after the 9 weeks intervention).
Population: Only participants who completed the Modified Conflict Tactics Scale-2 without missing data were included in the analysis. This explains why the number of participants analyzed is lower than the overall total number of study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KINDER Intervention
Number analyzed (Participants) | 31
score on a scale | -1.6 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of enrollment through 3 months post-enrollment.
Arm/Group | KINDER Intervention
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT05783102/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT05783102/ICF_001.pdf